CLINICAL TRIAL: NCT06599905
Title: Endogenous Pain Control Mechanisms Throughout the Migraine Cycle and in Chronic Migraine
Brief Title: Pain Control in Episodic and Chronic Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MigOA
Record Dates: First submitted 2024-07-11; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Migraine
Keywords: migraine; pain; offset analgesia; chronification
MeSH Terms: conditions — Migraine Disorders; Pain

STUDY DESIGN:
Intervention Model Description: To evaluate differences in the response to offset analgesia (OA) paradigm between episodic and chronic migraine patients and controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group with episodic migraine (EM) (Experimental): Subjects with episodic migraine (EM) with or without aura according to the International Headache Society (IHS) Classification (3rd edition).
  Interventions: Other: Chronic Migraine (CM)
- Group with chronic migraine (EC) (Experimental): Subjects with chronic migraine (CM) with or without Medication Overuse (MO) according to the International Headache Society (IHS) Classification (3rd edition).
  Interventions: Other: Episodic Migraine (EM)
- Control group (Other): Age- and sex-matched controls.
  Interventions: Other: Episodic Migraine (EM); Other: Chronic Migraine (CM)

INTERVENTIONS:
Other: Episodic Migraine (EM) — Three stimulus offset trials (OT) and three constant temperature trials (CT) applied to the forehead based on the individual heat pain threshold (HPT).
  Arms: Control group; Group with chronic migraine (EC)
Other: Chronic Migraine (CM) — Three stimulus offset trials (OT) and three constant temperature trials (CT) applied to the forehead based on the individual heat pain threshold (HPT).
  Arms: Control group; Group with episodic migraine (EM)

SUMMARY:
The phenomenon of offset analgesia (OA) refers to a disproportionately large decrease in perceived pain following a slight reduction in the intensity of a noxious heat stimulus. This phenomenon is considered as an indicator of the activation of the endogenous pain modulation system, whose dysfunction is implicated in the pathophysiology of migraine and other chronic pain conditions. This study aims to investigate pain processing mechanisms using the OA paradigm in individuals with episodic migraine (EM) during different phases of the migraine cycle and in those with chronic migraine (CM), with and without medication overuse headache (CMwoMOH and CM-MOH, respectively). A population of healthy subjects matched by sex and age will also be enrolled

DETAILED DESCRIPTION:
Migraine is a cyclic disorder marked by varying activity in different brain regions. It is generally believed that migraine involves a pronociceptive pain modulation pattern, likely due to impaired endogenous pain inhibitory systems. However, there are few studies in this respect, and different experimental approaches have produced mixed results, showing both normal and abnormal pain responses in migraine. Most research has focused only on episodic migraine (EM) during headache-free periods, leaving the role of pain modulation dysfunction in recurring migraines and the progression to chronic migraine unexplored. Conditioned Pain Modulation (CPM) tests, which measure the "pain inhibits pain" effect, are commonly used to assess inhibitory pain modulation. Studies comparing CPM responses in migraine sufferers and healthy individuals have yielded inconsistent findings, with some showing reduced inhibitory responses in migraineurs, while others found no difference. Offset Analgesia (OA) is another method used to study descending pain modulation systems in chronic pain conditions. Unlike CPM, OA examines temporal filtering of pain when dynamic noxious stimuli are applied and is characterized by a large reduction in pain sensation after a small decrease in a heat stimulus. Research indicates that central mechanisms, including the activation of descending pain modulatory and reward systems, play a significant role in OA. Only one study has explored the OA response in episodic migraine patients during headache-free intervals, finding no inhibitory pain modulation in the trigeminal area. This study aims to: 1) assess changes in pain modulation across the migraine cycle in EM patients, and 2) determine if different dysfunctional pain modulation patterns are present in chronic migraine, both with and without medication-overuse headache (CMwoMOH and CM-MOH).

Subjects and methods. The investigators will enroll 30 subjects with EM, 30 patients with CM (with and without MOH), and 30 healthy control subjects. Patients with EM during the preictal, ictal, and postictal phases will be also enrolled. All participants underwent an experimental paradigm consisting of three stimulus offset trials (OT) and three constant temperature trials (CT) applied to the forehead based on the individual heat pain threshold (HPT). All tests will be carried out by using a Q-sense CPM device (Medoc) and computerized visual analogue scale (CoVAS).

Experimental paradigms. All subjects will be assessed in a single experimental session. After obtaining written consent, participants will complete various questionnaires. The Heat Pain Threshold (HPT) will be then measured on the forehead (1st branch of the trigeminal nerve, V1), followed by three constant trials (CT) and three offset-analgesia trials (OT) in the same area. The following questionnaires will be administered: 12-item Allodynia Symptom Checklist (ASC-12), Migraine Disability Assessment (MIDAS), and Hospital Anxiety and Depression Scale (HADS).

ELIGIBILITY:
Inclusion Criteria:

* patients affected by episodic or chronic migraine according to the International Headache Society (IHS) Classification (3rd edition), aged 18 to 70 years

Exclusion Criteria:

* any other headache diagnosis according to the IHS classification
* other acute or chronic pain conditions
* serious internal, psychiatric, or neurological systemic diseases
* pregnancy, breastfeeding, skin pathologies in the tested trigeminal nerve area (V1)
* poor sleep quality the night before testing
* alcohol consumption or intense exercise within 24 hours prior to examination
* women were not assessed during their menstrual cycle.
* Use of migraine prophylactic medication for patients with EM.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Offset analgesia paradigm | Through study completion, an average of 2 years
  Differences in pain scores on the Visual Analog Scale and during the offset analgesia trial and the constant trials in patients with episodic migraine evaluated in the interictal period compared to patients with chronic migraine (with or without medication overuse) and healthy control subjects matched for sex and age

SECONDARY OUTCOMES:
Offset analgesia paradigm in different phase of episodic migraine | Through study completion, an average of 2 years
  Differences in pain scores on the Visual Analog Scale and during the offset analgesia trial and the constant trials in patients with episodic migraine evaluated in different phases of the migraine cycle (interictal, preictal, ictal, postictal).
Offset analgesia paradigm in chronic migraine with or without medication overuse headache | Through study completion, an average of 2 years
  Differences in pain scores on the Visual Analog Scale and during the offset analgesia trial and the constant trials in patients suffering from chronic migraine with or without medication overuse headache.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Cosentino, MD, Principal Investigator — Translational Neurophysiology - Headache and Neurorehabilitation Research Center
Locations (1):
- Clinical Trial Center, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cosentino G, Fierro B, Vigneri S, Talamanca S, Paladino P, Baschi R, Indovino S, Maccora S, Valentino F, Fileccia E, Giglia G, Brighina F. Cyclical changes of cortical excitability and metaplasticity in migraine: evidence from a repetitive transcranial magnetic stimulation study. Pain. 2014 Jun;155(6):1070-1078. doi: 10.1016/j.pain.2014.02.024. Epub 2014 Mar 13. PMID 24631596
- [Background] Schulte LH, May A. The migraine generator revisited: continuous scanning of the migraine cycle over 30 days and three spontaneous attacks. Brain. 2016 Jul;139(Pt 7):1987-93. doi: 10.1093/brain/aww097. Epub 2016 May 5. PMID 27190019
- [Background] Tassorelli C, Greco R, Silberstein SD. The endocannabinoid system in migraine: from bench to pharmacy and back. Curr Opin Neurol. 2019 Jun;32(3):405-412. doi: 10.1097/WCO.0000000000000688. PMID 30883435
- [Background] Szikszay TM, Adamczyk WM, Carvalho GF, May A, Luedtke K. Offset analgesia: somatotopic endogenous pain modulation in migraine. Pain. 2020 Mar;161(3):557-564. doi: 10.1097/j.pain.0000000000001739. PMID 31693545
- [Background] de Tommaso M, Losito L, Difruscolo O, Sardaro M, Libro G, Guido M, Lamberti P, Livrea P. Capsaicin failed in suppressing cortical processing of CO2 laser pain in migraine patients. Neurosci Lett. 2005 Aug 12-19;384(1-2):150-5. doi: 10.1016/j.neulet.2005.04.086. PMID 15927376
- [Background] de Tommaso M, Difruscolo O, Sardaro M, Libro G, Pecoraro C, Serpino C, Lamberti P, Livrea P. Effects of remote cutaneous pain on trigeminal laser-evoked potentials in migraine patients. J Headache Pain. 2007 Jun;8(3):167-74. doi: 10.1007/s10194-007-0385-8. Epub 2007 Jun 11. PMID 17563842
- [Background] Coppola G, Di Clemente L, Fumal A, Magis D, De Pasqua V, Pierelli F, Schoenen J. Inhibition of the nociceptive R2 blink reflex after supraorbital or index finger stimulation is normal in migraine without aura between attacks. Cephalalgia. 2007 Jul;27(7):803-8. doi: 10.1111/j.1468-2982.2007.01323.x. PMID 17598762
- [Background] Perrotta A, Serrao M, Sandrini G, Burstein R, Sances G, Rossi P, Bartolo M, Pierelli F, Nappi G. Sensitisation of spinal cord pain processing in medication overuse headache involves supraspinal pain control. Cephalalgia. 2010 Mar;30(3):272-84. doi: 10.1111/j.1468-2982.2009.01914.x. Epub 2010 Feb 15. PMID 19614707
- [Background] Grill JD, Coghill RC. Transient analgesia evoked by noxious stimulus offset. J Neurophysiol. 2002 Apr;87(4):2205-8. doi: 10.1152/jn.00730.2001. PMID 11929939
- [Background] Ligato D, Petersen KK, Morch CD, Arendt-Nielsen L. Offset analgesia: The role of peripheral and central mechanisms. Eur J Pain. 2018 Jan;22(1):142-149. doi: 10.1002/ejp.1110. Epub 2017 Sep 12. PMID 28898500